CLINICAL TRIAL: NCT05435287
Title: Critical Incident During Anaesthesia
Status: Completed | Type: Observational
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Kateryna Bielka, Associated professor at the Department of OF SURGERY, ANESTHESIOLOGY AND INTENSIVE THERAPY OF POSTGRADUATE EDUCATION, Bogomolets National Medical University
Other Study IDs: B77KL32iv5
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Critical Incident; Safety Issues
Keywords: patient safety; critical incident; anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A multicenter study in Ukrainian hospitals on compliance with the requirements for responding to critical cases in the operating room, and the availability of relevant documentation and checklists.

DETAILED DESCRIPTION:
Timely information and response to emergencies are important both in the context of patient safety and in the context of the hospital economy. The availability of information systems is one of the security requirements of the Helsinki Declaration of Patient Safety.

Ukraine has only just begun its path to implementing the Declaration of Helsinki in Ukrainian hospitals. The level of adherence to the recommendations can vary considerably depending on the region, the provision of the hospital and the effectiveness of the institution's internal management. In our survey of Ukrainian hospitals, only 74% of hospitals kept records of anaesthesia complications in general, with only 46% having separate electronic or paper documents to record complications; Also, the majority of respondent physicians (62.9%) reported the absence of checklists or algorithms for actions in case of emergencies or emergencies during anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* critical incident during anaesthesia: massive hemorrhage >1000ml, difficult intubation, severe hypotension, severe bradycardia, desaturation, cardiac arrest, high spinal block, anesthetic toxicity, miocardial ischemia, severe arhytmia etc

Exclusion Criteria:

* critical incidents without aneasthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, who had critical incident during anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Critical Incident During Anaesthesia | 5 months
  Critical Incident During Anaesthesia

SECONDARY OUTCOMES:
The use of the WHO Safe Surgery checklist | 5 months
  The use of the WHO Safe Surgery checklist
Keeping records of the critical incidents | 5 months
  Keeping records of the critical incidents during anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Iurii Kuchyn, PhD, Study Director — Bogomolets National Medical University
Locations (1):
- Bogomolets NMU, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu EH, Koh KF. A prospective audit of critical incidents in anaesthesia in a university teaching hospital. Ann Acad Med Singap. 2003 Nov;32(6):814-20. PMID 14716952
- [Background] Agbamu, P.O Et...al (2016) Critical Incidents and Near Misses During Anaesthesia: a Prospective Audit.13th Annual Scientific, Conference and Gathering Held at College of Medicine, University of Lagos, Idi Araba.
- [Background] Amucheazi AO, Ajuzieogu OV. Critical incidents during anesthesia in a developing country: A retrospective audit. Anesth Essays Res. 2010 Jul-Dec;4(2):64-8. doi: 10.4103/0259-1162.73508. PMID 25885231
- [Background] Ahluwalia J, Marriott L. Critical incident reporting systems. Semin Fetal Neonatal Med. 2005 Feb;10(1):31-7. doi: 10.1016/j.siny.2004.09.012. PMID 15698968
- [Derived] Bielka K, Kuchyn I, Frank M, Sirenko I, Yurovich A, Slipukha D, Lisnyy I, Soliaryk S, Posternak G. Critical incidents during anesthesia: prospective audit. BMC Anesthesiol. 2023 Jun 14;23(1):206. doi: 10.1186/s12871-023-02171-4. PMID 37316789